CLINICAL TRIAL: NCT04011059
Title: Randomized Study as Proof of Concept of Coronary Revascularization Surgery With Injection of Wharton's Jelly-derived Mesenchymal Cells and Placement of an Epicardial Extracellular Matrix Patch Seeded With WJ-MSCs in Patients With Ischemic Cardiomyopathy
Brief Title: Randomized Study of Coronary Revascularization Surgery With Injection of WJ-MSCs and Placement of an Epicardial Extracellular Matrix
Acronym: scorem-cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital San Vicente Fundación (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government); IPS Universitaria Servicios de Salud Universidad de Antioquia (Unknown); Hospital San Vicente Fundación - Rionegro (Unknown)
Responsible Party: Principal Investigator, Luis Horacio Atehortua Lopez, Clinical Professor, Hospital San Vicente Fundación
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2019-06-15; First posted 2019-07-08 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Diseases; Heart Failure; Coronary Artery Disease; Mesenchymal Stem Cell Transplantation; Regenerative Medicine
Keywords: Heart Failure; Cardiomyopathies; Coronary Artery Disease; Ischemic Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Coronary Artery Disease; Cardiomyopathies

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be conducted as a proof of concept in 40 patients with previous myocardial infarction and a viable myocardial zone with indications for coronary artery bypass grafts. Twenty patients will be included in each treatment arm over 36 months. One group will undergo revascularization surgery, extracellular matrix patch placement and injection of cell culture medium; the other group will undergo revascularization surgery, extracellular matrix patch placement on the epicardial surface with cultured WJ-MSCs and injection of WJ-MSCs around the infarcted zone.
  The allocation of treatments will be defined by block sizes of 2, 4 and 6, randomly determined by a random number generator (ralloc, Stata Co. 8,2). This assignment will only be known by the tissue bank that will deliver the syringes with the solution to be administered and the epicardium patches to the study participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This assignment will only be known by the tissue bank that will deliver the syringes with the solution to be administered and the epicardium patches to the study participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison/control group (Placebo Comparator): Revascularization surgery, placement of an extracellular matrix patch without WJ-MSCs and injection of culture medium without WJ-MSCs will be performed.
  Interventions: Biological: Wharton's jelly-derived mesenchymal cells
- Experimental group (Active Comparator): Revascularization surgery, placement of an extracellular matrix patch with WJ-MSCs cultured on the epicardial surface and injection of WJ-MSCs around the infarcted zone will be performed.
  Interventions: Biological: Wharton's jelly-derived mesenchymal cells

INTERVENTIONS:
Biological: Wharton's jelly-derived mesenchymal cells — Revascularization surgery, placement of an extracellular matrix patch with WJ-MSCs cultured on the epicardial surface and injection of WJ-MSC around the infarcted zone.

SUMMARY:
Ischemic heart disease is one of the most important causes of mortality and morbidity in the Western world and is a public health problem. Among ischemic heart diseases, myocardial infarction has specific significance because the cardiac muscle does not have sufficient and adequate capacity to regenerate; therefore, necrosis of a region leads to the formation of a fibrous scar. Infarction can lead to a progressive and irreversible decrease in cardiac function, resulting in heart failure (HF) syndrome, depending on the area affected by this scar, via a ventricular remodeling mechanism.

In recent years, HF has been revealed as a major public health problem due to its incidence and its social, economic and especially human impact, as it represents a serious limitation of the quality of life of individuals. The prevalence of HF in the general population of the United States and the United Kingdom is approximately 1%, and in those older than 75 years, the prevalence varies between 5 and 10%. Regarding its prognosis, recent data from the Framingham Study indicate that at 5 years, the mortality rate of HF is 75% in men and 62% in women; the mean mortality rate of all cancers is 50%.

The molecular basis of congestive HF is the absence of cardiac cells capable of regenerating the heart muscle. Despite the publication of recent studies suggesting the existence of stem cells capable of regenerating cardiomyocytes destroyed because of myocardial infarction, in humans, the capacity of these cells is insufficient to replace the cells destroyed due to necrosis secondary to ischemia.

In recent years, the accumulation of results derived from preclinical studies has allowed the development of the first clinical trials of the feasibility and safety of cardiac regeneration using cellular therapy. Several studies have shown that t cells exist in adult bone marrow, such as mesenchymal stem cells, hematopoietic stem cells and, more recently, multipotent stem cells (MAPC), with the ability to differentiate into endothelial tissue and cardiac muscle, which can contribute to the regeneration of damaged myocardial tissue and improve cardiac function in animal infarction models. However, cell therapy research has moved rapidly toward the use of more undifferentiated cells rather than hematopoietic lineages, such as mesenchymal cells. These cells can be obtained from different sources, with a tendency toward the use of characterized allogeneic cells, which are immediately available in the potential recipient. Given that this type of therapy has not been rigorously investigated in Latin America, we aim to determine the effect of therapy using Wharton's jelly-derived mesenchymal cells (WJ-MSCs) from the human umbilical cord on neomyogenesis in patients with previous myocardial infarction who are undergoing open revascularization. Our hospital has some experience with regenerative therapy, both in patients with acute myocardial infarction and chronic infarction, with encouraging results that support this new phase of inter-institutional research.

Objective: To evaluate the safety and estimate the effect of coronary revascularization accompanied by intramyocardial injection of WJ-MSCs and the placement of an extracellular matrix patch seeded with WJ-MSCs compared to coronary revascularization accompanied by injection of culture medium without the presence of WJ-MSC and placement of an extracellular matrix patch without seeding with WJ-MSC on global and regional cardiac function, myocardial viability and the incidence of adverse effects determined as ventricular arrhythmias.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted as a proof of concept in 40 patients with previous myocardial infarction and a viable myocardial zone with indications for coronary artery bypass grafts. Twenty patients will be included in each treatment arm over 36 months. One group will undergo revascularization surgery, extracellular matrix patch placement and injection of cell culture medium; the other group will undergo revascularization surgery, extracellular matrix patch placement on the epicardial surface with cultured WJ-MSCs and injection of WJ-MSCs around the infarcted zone.

The allocation of treatments will be defined by block sizes of 2, 4 and 6, randomly determined by a random number generator (ralloc, Stata Co. 8,2). This assignment will only be known by the tissue bank that will deliver the syringes with the solution to be administered and the epicardium patches to the study participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of coronary disease, performed by coronary angiography, requiring conventional coronary revascularization surgery
* History of myocardial infarction; evidence of akinesia or regional dyskinesia more than 1 week old
* Ejection fraction less than 40%
* Age between 30 and 75 years
* Negative serology for HIV, hepatitis B virus (HBV), and hepatitis C virus HCV
* Negative pregnancy test for women of childbearing age
* Patients who sign the informed consent complying with all of the provisions of current regulations in Colombia

Exclusion Criteria:

* History of myocardial infarction with ST-segment elevation within 2 weeks prior to surgery
* History of myocardial infarction without ST-segment elevation within the previous week (the decision to include these patients within the first week after suffering a non-ST elevation infarction is at the discretion of the research team)
* Previous history of tachycardia or ventricular fibrillation
* History of active neoplasia or previous chemotherapy treatment
* Severe or uncontrolled concomitant disease (i.e., poorly controlled chronic kidney or liver failure)
* Patients who, due to their place of residence, mental health or social situation, have difficulty meeting the conditions of the protocol
* Women who are pregnant or breast-feeding
* Patients or legal representatives withdrawing informed consent at any time during the study.
* Previous history of heart transplant
* Patients with functional organ impairment: liver function: total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase greater than 2 times the upper reference limit; kidney function: serum creatinine > 1.5 mg/dl or creatinine clearance < 60 ml/min.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-02 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | 12 months
  Percentage of improvement in left ventricular ejection fraction (LVEF) on transthoracic echocardiography and cardiac magnetic resonance imaging (MRI)
Final diastolic and systolic volumes | 12 months
  Percentage of improvement of the final diastolic and systolic volumes on transthoracic echocardiography and cardiac MRI
Left ventricule viability | 12 months
  Effect on viability, defined as a percentage of wall involvement, and improvement in segment-to-segment contractility measured with MRI
Ventricular arrhythmias | 12 months
  Incidence of ventricular arrhythmias defined as nonsustained ventricular tachycardia (NSTV) or high- or low-grade ventricular extrasystoles

SECONDARY OUTCOMES:
Estimated functional status | 12 months
  Recovery of the estimated functional status according to the New York Heart Association (NYHA) classification
Change in the median score of Quality of life | 12 months
  Change in the median score for quality of life of the Minnesota Living with Heart Failure Questionnaire (MLHFQ)
Delayed enhancement of the left ventricle | 12 months
  Changes in the delayed enhancement of the left ventricle on MRI, defined as percentage of the wall thickness involved when adding each segment visually
Improvement in the 6-minute walk test | 12 months
  Improvement in the 6-minute walk test, defined as the percentage of change of the distance traveled
Mortality at 3 and 12 months due to cardiovascular causes | 12 months
  Mortality at 3 and 12 months due to cardiovascular causes
Mortality at 3 and 12 months due to all causes | 12 months
  Mortality at 3 and 12 months due to all causes

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital San Vicente Fundación, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher SA, Doree C, Mathur A, Martin-Rendon E. Meta-analysis of cell therapy trials for patients with heart failure. Circ Res. 2015 Apr 10;116(8):1361-77. doi: 10.1161/CIRCRESAHA.116.304386. Epub 2015 Jan 28. PMID 25632038
- [Background] Velásquez Ó, Senior JM, Cuéllar F, Velásquez M, García LF, Navas C, et al. Autologous intramyocardial transplant of bone marrow derived stem cells for revascularization in ischemic chronic cardiopathy. Rev Col Cardiol [Internet]. 2005 [cited 2018 May 12];12(12):120-5633.
- [Background] Gómez E. Chapter 2. Introducción, epidemiología de la falla cardiaca e historia de las clínicas de falla cardiaca en Colombia. Rev Colomb Cardiol [Internet]. 2016 Mar 1 [cited 2018 May 12];23:6-12.
- [Background] Cowie MR, Mosterd A, Wood DA, Deckers JW, Poole-Wilson PA, Sutton GC, Grobbee DE. The epidemiology of heart failure. Eur Heart J. 1997 Feb;18(2):208-25. doi: 10.1093/oxfordjournals.eurheartj.a015223. No abstract available. PMID 9043837
- [Background] Trainini JC, Herreros J, Coto E otero, Aguilar JC. La "duda clave" de Torrent Guasp. Cirugía Cardiovasc [Internet]. 2011;18(2):77-81
- [Background] Wang WE, Li L, Xia X, Fu W, Liao Q, Lan C, Yang D, Chen H, Yue R, Zeng C, Zhou L, Zhou B, Duan DD, Chen X, Houser SR, Zeng C. Dedifferentiation, Proliferation, and Redifferentiation of Adult Mammalian Cardiomyocytes After Ischemic Injury. Circulation. 2017 Aug 29;136(9):834-848. doi: 10.1161/CIRCULATIONAHA.116.024307. Epub 2017 Jun 22. PMID 28642276
- [Background] Garbern JC, Lee RT. Cardiac stem cell therapy and the promise of heart regeneration. Cell Stem Cell. 2013 Jun 6;12(6):689-98. doi: 10.1016/j.stem.2013.05.008. PMID 23746978
- [Background] Hong KU, Bolli R. Cardiac stem cell therapy for cardiac repair. Curr Treat Options Cardiovasc Med. 2014 Jul;16(7):324. doi: 10.1007/s11936-014-0324-3. PMID 24903489
- [Background] Zwetsloot PP, Vegh AM, Jansen of Lorkeers SJ, van Hout GP, Currie GL, Sena ES, Gremmels H, Buikema JW, Goumans MJ, Macleod MR, Doevendans PA, Chamuleau SA, Sluijter JP. Cardiac Stem Cell Treatment in Myocardial Infarction: A Systematic Review and Meta-Analysis of Preclinical Studies. Circ Res. 2016 Apr 15;118(8):1223-32. doi: 10.1161/CIRCRESAHA.115.307676. Epub 2016 Feb 17. PMID 26888636
- [Background] Menasche P, Hagege AA, Vilquin JT, Desnos M, Abergel E, Pouzet B, Bel A, Sarateanu S, Scorsin M, Schwartz K, Bruneval P, Benbunan M, Marolleau JP, Duboc D. Autologous skeletal myoblast transplantation for severe postinfarction left ventricular dysfunction. J Am Coll Cardiol. 2003 Apr 2;41(7):1078-83. doi: 10.1016/s0735-1097(03)00092-5. PMID 12679204
- [Background] Patel AN, Geffner L, Vina RF, Saslavsky J, Urschel HC Jr, Kormos R, Benetti F. Surgical treatment for congestive heart failure with autologous adult stem cell transplantation: a prospective randomized study. J Thorac Cardiovasc Surg. 2005 Dec;130(6):1631-8. doi: 10.1016/j.jtcvs.2005.07.056. Epub 2005 Oct 26. PMID 16308009
- [Background] American College of Cardiology. K, Malliaras K, Shen D, Tseliou E, Ionta V, Smith J, et al. Journal of the American College of Cardiology. [Internet]. Vol. 59, Journal of the American College of Cardiology. Elsevier Biomedical; 1983 [cited 2018 May 12]. 256-264
- [Background] Tompkins BA, Balkan W, Winkler J, Gyongyosi M, Goliasch G, Fernandez-Aviles F, Hare JM. Preclinical Studies of Stem Cell Therapy for Heart Disease. Circ Res. 2018 Mar 30;122(7):1006-1020. doi: 10.1161/CIRCRESAHA.117.312486. PMID 29599277
- [Background] Caplan AI. All MSCs are pericytes? Cell Stem Cell. 2008 Sep 11;3(3):229-30. doi: 10.1016/j.stem.2008.08.008. No abstract available. PMID 18786406
- [Background] Caplan AI. Adult mesenchymal stem cells for tissue engineering versus regenerative medicine. J Cell Physiol. 2007 Nov;213(2):341-7. doi: 10.1002/jcp.21200. PMID 17620285
- [Background] Caplan AI. Review: mesenchymal stem cells: cell-based reconstructive therapy in orthopedics. Tissue Eng. 2005 Jul-Aug;11(7-8):1198-211. doi: 10.1089/ten.2005.11.1198. PMID 16144456
- [Background] Barminko J, Gray A, Maguire T, Schloss R, Yarmush ML. Mesenchymal Stem Cell Therapy. Mesenchymal Stem Cell Therapy. 405-421, 2013
- [Background] Wolfe M, Pochampally R, Swaney W, Reger RL. Isolation and culture of bone marrow-derived human multipotent stromal cells (hMSCs). Methods Mol Biol. 2008;449:3-25. doi: 10.1007/978-1-60327-169-1_1. PMID 18370080
- [Background] Tanavde V, Vemuri MC. Mesenchymal stromal cells in the clinic: What do the clinical trials say? In: Mesenchymal Stem Cell Therapy. 423-33, 2013
- [Background] Wang HS, Hung SC, Peng ST, Huang CC, Wei HM, Guo YJ, Fu YS, Lai MC, Chen CC. Mesenchymal stem cells in the Wharton's jelly of the human umbilical cord. Stem Cells. 2004;22(7):1330-7. doi: 10.1634/stemcells.2004-0013. PMID 15579650
- [Background] Weiss ML, Anderson C, Medicetty S, Seshareddy KB, Weiss RJ, VanderWerff I, Troyer D, McIntosh KR. Immune properties of human umbilical cord Wharton's jelly-derived cells. Stem Cells. 2008 Nov;26(11):2865-74. doi: 10.1634/stemcells.2007-1028. Epub 2008 Aug 14. PMID 18703664
- [Background] Bensaid W, Triffitt JT, Blanchat C, Oudina K, Sedel L, Petite H. A biodegradable fibrin scaffold for mesenchymal stem cell transplantation. Biomaterials. 2003 Jun;24(14):2497-502. doi: 10.1016/s0142-9612(02)00618-x. PMID 12695076
- [Background] Baraniak PR, McDevitt TC. Scaffold-free culture of mesenchymal stem cell spheroids in suspension preserves multilineage potential. Cell Tissue Res. 2012 Mar;347(3):701-11. doi: 10.1007/s00441-011-1215-5. Epub 2011 Aug 11. PMID 21833761
- [Background] Timmers L, Lim SK, Hoefer IE, Arslan F, Lai RC, van Oorschot AA, Goumans MJ, Strijder C, Sze SK, Choo A, Piek JJ, Doevendans PA, Pasterkamp G, de Kleijn DP. Human mesenchymal stem cell-conditioned medium improves cardiac function following myocardial infarction. Stem Cell Res. 2011 May;6(3):206-14. doi: 10.1016/j.scr.2011.01.001. Epub 2011 Jan 28. PMID 21419744
- [Background] Chong JJ, Chandrakanthan V, Xaymardan M, Asli NS, Li J, Ahmed I, Heffernan C, Menon MK, Scarlett CJ, Rashidianfar A, Biben C, Zoellner H, Colvin EK, Pimanda JE, Biankin AV, Zhou B, Pu WT, Prall OW, Harvey RP. Adult cardiac-resident MSC-like stem cells with a proepicardial origin. Cell Stem Cell. 2011 Dec 2;9(6):527-40. doi: 10.1016/j.stem.2011.10.002. PMID 22136928
- [Background] Singh A, Singh A, Sen D. Mesenchymal stem cells in cardiac regeneration: a detailed progress report of the last 6 years (2010-2015). Stem Cell Res Ther. 2016 Jun 4;7(1):82. doi: 10.1186/s13287-016-0341-0. PMID 27259550
- [Background] Beltrami AP, Urbanek K, Kajstura J, Yan SM, Finato N, Bussani R, Nadal-Ginard B, Silvestri F, Leri A, Beltrami CA, Anversa P. Evidence that human cardiac myocytes divide after myocardial infarction. N Engl J Med. 2001 Jun 7;344(23):1750-7. doi: 10.1056/NEJM200106073442303. PMID 11396441
- [Background] Ghostine S, Carrion C, Souza LC, Richard P, Bruneval P, Vilquin JT, Pouzet B, Schwartz K, Menasche P, Hagege AA. Long-term efficacy of myoblast transplantation on regional structure and function after myocardial infarction. Circulation. 2002 Sep 24;106(12 Suppl 1):I131-6. PMID 12354722
- [Background] Dominici M, Le Blanc K, Mueller I, Slaper-Cortenbach I, Marini F, Krause D, Deans R, Keating A, Prockop Dj, Horwitz E. Minimal criteria for defining multipotent mesenchymal stromal cells. The International Society for Cellular Therapy position statement. Cytotherapy. 2006;8(4):315-7. doi: 10.1080/14653240600855905. PMID 16923606
- [Background] Brooke G, Cook M, Blair C, Han R, Heazlewood C, Jones B, Kambouris M, Kollar K, McTaggart S, Pelekanos R, Rice A, Rossetti T, Atkinson K. Therapeutic applications of mesenchymal stromal cells. Semin Cell Dev Biol. 2007 Dec;18(6):846-58. doi: 10.1016/j.semcdb.2007.09.012. Epub 2007 Sep 18. PMID 18024097
- [Background] Keating A. Mesenchymal stromal cells. Curr Opin Hematol. 2006 Nov;13(6):419-25. doi: 10.1097/01.moh.0000245697.54887.6f. PMID 17053453
- [Background] Chen PM, Yen ML, Liu KJ, Sytwu HK, Yen BL. Immunomodulatory properties of human adult and fetal multipotent mesenchymal stem cells. J Biomed Sci. 2011 Jul 18;18(1):49. doi: 10.1186/1423-0127-18-49. PMID 21762539
- [Background] Lalu MM, McIntyre L, Pugliese C, Fergusson D, Winston BW, Marshall JC, Granton J, Stewart DJ; Canadian Critical Care Trials Group. Safety of cell therapy with mesenchymal stromal cells (SafeCell): a systematic review and meta-analysis of clinical trials. PLoS One. 2012;7(10):e47559. doi: 10.1371/journal.pone.0047559. Epub 2012 Oct 25. PMID 23133515
- [Background] Lai RC, Yeo RWY, Tan SS, Zhang B, Yin Y, Sze NSK, et al. Mesenchymal stem cell exosomes: The future MSC-based therapy? In: Mesenchymal Stem Cell Therapy. 39-61, 2013
- [Background] Barminko J, Gray A, Maguire T, Schloss R, Yarmush ML. Mesenchymal stromal cell mechanisms of immunomodulation and homing. In: Mesenchymal Stem Cell Therapy. 15-38, 2013.
- [Background] Gaafar T, Attia W, Mahmoud S, Sabry D, Aziz OA, Rasheed D, Hamza H. Cardioprotective Effects of Wharton Jelly Derived Mesenchymal Stem Cell Transplantation in a Rodent Model of Myocardial Injury. Int J Stem Cells. 2017 May 30;10(1):48-59. doi: 10.15283/ijsc16063. PMID 28446005
- [Background] Rabbani S, Soleimani M, Imani M, Sahebjam M, Ghiaseddin A, Nassiri SM, Majd Ardakani J, Tajik Rostami M, Jalali A, Mousanassab B, Kheradmandi M, Ahmadi Tafti SH. Regenerating Heart Using a Novel Compound and Human Wharton Jelly Mesenchymal Stem Cells. Arch Med Res. 2017 Apr;48(3):228-237. doi: 10.1016/j.arcmed.2017.03.019. PMID 28923324
- [Background] Balbi C, Bollini S. Fetal and perinatal stem cells in cardiac regeneration: Moving forward to the paracrine era. Placenta. 2017 Nov;59:96-106. doi: 10.1016/j.placenta.2017.04.008. Epub 2017 Apr 12. PMID 28416208
- [Background] Nimsanor N, Phetfong J, Plabplueng C, Jangpatarapongsa K, Prachayasittikul V, Supokawej A. Inhibitory effect of oxidative damage on cardiomyocyte differentiation from Wharton's jelly-derived mesenchymal stem cells. Exp Ther Med. 2017 Dec;14(6):5329-5338. doi: 10.3892/etm.2017.5249. Epub 2017 Oct 2. PMID 29285060
- [Background] Munir H, Luu NT, Clarke LS, Nash GB, McGettrick HM. Comparative Ability of Mesenchymal Stromal Cells from Different Tissues to Limit Neutrophil Recruitment to Inflamed Endothelium. PLoS One. 2016 May 12;11(5):e0155161. doi: 10.1371/journal.pone.0155161. eCollection 2016. PMID 27171357